CLINICAL TRIAL: NCT06577597
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Safety, Tolerability and Pharmacokinetics of Single Doses of GSK3923868 Administered Via Dry Powder Inhaler to Healthy Participants of Chinese, Japanese and European Ancestry
Brief Title: Safety, Tolerability and Blood Sampling of GSK3923868 Administered Via Dry Powder Inhaler to Healthy Participants of Chinese, Japanese and European Ancestry
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 218320
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Tract Infections
Keywords: GSK3923868; Safety; Tolerability; Pharmacokinetics; Healthy participants; Phosphatidylinositol 4-kinase beta (PI4KB)
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blinded study where participants and site staff will be blinded to the study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSK3923868 (Experimental): Participants from Chinese, Japanese and European ancestries will receive single dose of GSK3923868.
  Interventions: Drug: GSK3923868
- Placebo (Placebo Comparator): Participants from Chinese, Japanese and European ancestries will receive single dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3923868 — Participants will receive single dose of GSK3923868.
  Arms: GSK3923868
Drug: Placebo — Participants will receive single dose of Placebo.
  Arms: Placebo

SUMMARY:
This study is designed to understand how the drug GSK3923868 works in the bodies of healthy people from Japanese, Chinese, and European ancestries. This is important to meet the rules for including these groups in future worldwide studies. The study is carefully planned to reduce differences that might come from comparing results across different studies and locations, making it easier to compare results between these ethnic groups. The main goal is to check if GSK3923868 is safe and easy to tolerate when given as a single inhaled dose to healthy people from these three ancestries. The study also wants to see how the drug moves in the blood after a single inhaled dose in these groups. On the first day of the study, participants will be randomly chosen to receive either a single dose of GSK3923868 or a placebo. The aim is to have enough people take part so that 10 healthy people from each ancestry group (a total of 30 people) can successfully finish the study. Should a participant withdraw from the study before completion, the GSK Medical Monitor and the investigator may select a replacement. The replacement participant will be assigned the same treatment as the original participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are generally healthy as determined by medical evaluation based on screening medical history, physical examination, vital signs, electrocardiogram (ECG) assessment, pulmonary function testing and laboratory tests
* Body weight at least 50.0 kilograms (kg) for male participants or at least 45.0 kg for female participants
* Body Mass Index (BMI) within the range of 18.0-28.0 kilograms per square meter (kg/m^2) (inclusive)
* A female participant is eligible to participate if she is not pregnant or breastfeeding and is a Woman of non-childbearing potential (WONCBP); or Woman of childbearing potential (WOCBP) and using an acceptable contraceptive method; or A WOCBP must have a negative highly sensitive pregnancy test within 30 days before the first dose of study intervention
* Informed consent: Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Participants of Chinese ancestry are eligible if they are born in mainland China, Hong Kong or Taiwan; descendant of 4 ethnic Chinese grandparents and 2 ethnic Chinese parents; have lived outside mainland China, Hong Kong or Taiwan for less than 10 years at the time of screening
* Participants of Japanese ancestry are eligible if they are born in Japan, descendent of 4 ethnic Japanese grandparents and 2 ethnic Japanese parents; have lived outside Japan less than 10 years at the time of screening
* Participants of European ancestry are eligible if they self-identified as being European ancestry (that is, from the original people of Europe) irrespective of place of birth and current place of residence; descendent of 4 grandparents and 2 parents of European ancestry

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data
* Serum Alanine transaminase (ALT) and Aspartate Aminotransferase (AST) above Upper limit of normal (ULN)
* Total Bilirubin above ULN (isolated bilirubin above ULN is acceptable if total bilirubin is fractionated and direct bilirubin less than [<] 35 percent [%])
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QTcF greater than (>) 450 milliseconds (msec) at Screening visit based on the average of triplicate ECGs
* Past or intended use of over-the-counter or prescription medication, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the first dose of study treatment, unless in the opinion of the investigator and the GSK Medical Monitor (if necessary), the medication will not interfere with the study procedures or compromise participant safety
* Recent donation of blood or blood products such that participation in this study would result in loss of blood in excess of 500 mL within a 60-day period.
* Exposure to more than 4 new chemical or molecular entities within 12 months before the first dosing day
* Current enrolment or past participation in a clinical trial and has received an investigational product within the following time period before the first dosing day in this study: 45 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* FEV1 <80% predicted normal value at Screening
* Presence of hepatitis B surface antigen at screening or within 3 months prior to first dose of study intervention
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention
* Positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention
* Positive pre-study drug/alcohol screen
* Positive HIV antibody test
* Current or history of drug abuse
* Current or previous use of tobacco- or nicotine-containing products (e.g. cigarettes, nicotine patches or electronic devices) within 6 months before screening and/or have a smoking pack history of >5 pack years
* Positive urine cotinine test indicative of recent smoking at Screening or admission to the clinical research unit
* History of regular alcohol consumption within 6 months prior to the study defined as: An average weekly intake of >14 units for males and females
* Sensitivity to the study intervention or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse events (AE) | Up to Day 14 (End of follow up)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention
Number of Participants with Serious Adverse events (SAE) | Up to Day 14 (End of follow up)
  An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in the offspring of a study participant; abnormal pregnancy outcome; or is a suspected transmission of any infectious agent via an authorized medicinal product.
Number of Participants with Clinically Significant Changes in Laboratory Values | Up to Day 14 (End of follow up)
  Clinically significant changes in laboratory values (Clinical Chemistry, Haematology and Coagulation Clinical Chemistry, Haematology, and Coagulation) will be assessed.
Number of Participants with Clinically Significant Changes in Laboratory values | Up to Day 14 (End of follow up)
  Clinically significant changes in Laboratory values (Urinalysis) will be assessed.
Number of Participants with Clinically Significant Changes in Vital signs | Up to Day 14 (End of follow up)
  Clinically significant changes in Vital signs (systolic and diastolic blood pressure, heart rate, respiration rate, pulse oximetry and oral temperature) will be assessed.
Number of Participants with Clinically Significant Changes in 12-lead Electrocardiogram (ECG) | Up to Day 14 (End of follow up)
  Clinically significant changes in 12-lead ECG will be assessed.
Number of Participants with Clinically Significant Changes in Spirometry Measurements | On Day 14 (End of follow up)
  Number of participants with clinically significant changes in Spirometry measurements.
Area Under the Plasma GSK3923868 Concentration Versus Time Curve from Time Zero to Last Quantifiable Concentration (AUC[0-t]) of GSK3923868 | Up to Day 4
  Blood samples will be collected at the specified timepoints for the pharmacokinetics (PK) assessments.
Area under the Plasma GSK3923868 Concentration versus Time Curve from Time zero to Infinity (AUC[0-inf]) of GSK3923868 | Up to Day 4
  Blood samples will be collected at the specified timepoints for the PK assessments.
Maximum Observed GSK3923868 Plasma Concentration (Cmax) of GSK3923868 | Up to Day 4
  Blood samples will be collected at the specified timepoints for the PK assessments.
Time to Maximum Observed Plasma Drug Concentration (Tmax) of GSK3923868 | Up to Day 4
  Blood samples will be collected at the specified timepoints for the PK assessments.
Terminal Half-life (T1/2) of GSK3923868 | Up to Day 4
  Blood samples will be collected at the specified timepoints for the PK assessments.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/